CLINICAL TRIAL: NCT04617483
Title: A Randomized, Double-Blinded Clinical Trial, to Evaluate the Non-inferiority of the Commercial Scale Inactivated SARS-CoV-2 Vaccine Against That of the Pilot Scale Among Adults Aged 26-45 Years, and the Open-labelled, Bridging Non-inferiority of the Vaccine Induced Immunogenicity in Elderly Against That in Adults
Brief Title: Study of the Commercial Scale SARS-CoV-2 Vaccine Against the Pilot Scale Among Adults, and Bridging Study of the Immunogenicity in Elderly Against That in Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sinovac Research and Development Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Sinovac Biotech Co., Ltd (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PRO-nCOV-3001
Record Dates: First submitted 2020-11-04; First posted 2020-11-05 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2020-11

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — Aging

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The first part of the study is a double-blinded trial, the second part is a open-label research.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Aged 26-45, Commercial Scale (Experimental): Commercial scale inactivated SARS-CoV-2 vaccine in adults aged 26-45 years.
  Interventions: Biological: Two doses of commercial scale inactivated SARS-CoV-2 vaccine at the schedule of day 0,14
- Aged 18-59, Pilot Scale (Experimental): Pilot scale inactivated SARS-CoV-2 vaccine in adults aged 18-59 years.
  Interventions: Biological: Two doses of pilot scale inactivated SARS-CoV-2 vaccine at the schedule of day 0,14
- Aged ≥60, Pilot Scale (Experimental): Pilot scale inactivated SARS-CoV-2 vaccine in elderly aged above 60 years.
  Interventions: Biological: Two doses of pilot scale inactivated SARS-CoV-2 vaccine at the schedule of day 0,14 in elderly

INTERVENTIONS:
Biological: Two doses of commercial scale inactivated SARS-CoV-2 vaccine at the schedule of day 0,14 — The antigen content of the commercial scale inactivated SARS-CoV-2 vaccine was 600SU/0.5ml, vaccinated in the age group 26-45.
  Arms: Aged 26-45, Commercial Scale
Biological: Two doses of pilot scale inactivated SARS-CoV-2 vaccine at the schedule of day 0,14 — The antigen content of the pilot scale inactivated SARS-CoV-2 vaccine was 600SU/0.5ml, vaccinated in the age group 18-59.
  Arms: Aged 18-59, Pilot Scale
Biological: Two doses of pilot scale inactivated SARS-CoV-2 vaccine at the schedule of day 0,14 in elderly — The antigen content of the pilot scale inactivated SARS-CoV-2 vaccine was 600SU/0.5ml, vaccinated in the age group above 60.
  Arms: Aged ≥60, Pilot Scale

SUMMARY:
This study is a randomized, double-blinded clinical Trial, to evaluate the non-inferiority of the commercial scale Inactivated SARS-CoV-2 vaccine against that of the pilot scale among adults aged 26-45 years, and the open-labelled, bridging non-inferiority of the vaccine induced immunogenicity in elderly against that in adults.

DETAILED DESCRIPTION:
This study is a randomized, double-blinded clinical Trial, to evaluate the non-inferiority of the commercial scale Inactivated SARS-CoV-2 vaccine against that of the pilot scale among adults aged 26-45 years, and the open-labelled, bridging non-inferiority of the vaccine induced immunogenicity in elderly against that in adults. The experimental vaccine was manufactured by Sinovac Research & Development Co.,Ltd. Totally 1040 subjects，including: 130 subjects aged 18~25 years; 520 subjects aged 26~45 years, with 260 in each group; 130 subjects aged 46~59 years; 260 subjects aged ≥60 years.

Subjects will be assigned to receive two doses of medium-dosage vaccine on the schedule of 0,14.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults aged 18-59 or elderly aged ≥60 years;
2. Proven legal identity.

Exclusion Criteria:

1. Travel/residence history of communities with reported cases within 14 days before trial;
2. History of exposure to Novel Coronavirus infection (nucleic acid positive) within 14 days prior to the trial;
3. Exposed to patients with fever or respiratory symptoms from communities with reported cases within 14 days prior to the trial;
4. Two or more cases of fever and/or respiratory symptoms in a small area such as home, office, school and class within 14 days prior to the trial;
5. History of SARS-CoV-2 infection;
6. History of asthma, history of allergy to vaccines or vaccine ingredients, and severe adverse reactions to vaccines, such as urticaria, dyspnea, and angioneurotic edema;
7. Congenital malformations or developmental disorders, genetic defects, severe malnutrition, etc.;
8. Autoimmune disease or immunodeficiency/immunosuppression;
9. Patients with serious chronic diseases, serious cardiovascular diseases, uncontrolled hypertension and diabetes, liver and kidney diseases, malignant tumors, etc.;
10. Serious neurological disorder (epilepsy, convulsions or convulsions) or psychosis;
11. History of thyroid disease or thyroidectomy, absence of spleen, functional absence of spleen, and absence of spleen or splenectomy caused by any circumstance;
12. Coagulation dysfunction (such as coagulation factor deficiency, coagulation disease, platelet abnormality) or obvious bruising or coagulation disorder diagnosed by doctors;
13. Immunosuppressive therapy, cytotoxic therapy, inhaled corticosteroids (excluding corticosteroid spray therapy for allergic rhinitis, and surface corticosteroid therapy for acute non-complicated dermatitis) in the past 6 months;
14. Long history of alcohol or drug abuse;
15. Received blood products within 3 months prior to receiving the vaccine;
16. Received other research drugs within 30 days prior to receiving the vaccine;
17. Received live attenuated vaccine within 14 days prior to receiving the vaccine;
18. Received subunit or inactivated vaccine within 7 days prior to receiving the vaccine;
19. Onset of various acute or chronic diseases within 7 days prior to the study;
20. Axillary temperature of >37.0℃ before inoculation of the vaccine;
21. Those who are already pregnant (including a positive urine pregnancy test) or are breastfeeding, planning to become pregnant within 2 months;
22. In the opinion of the investigator, the participants had any other factors that made them unsuitable to participate in the clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1040 (Actual)
Dates: Start 2020-10-31 (Actual); Primary Completion 2020-11-28 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Immunogenicity index-geometric mean titer(GMT) of neutralizing antibody | Day 14 after the full course vaccination
  Neutralizing antibody assay will be performed using the micro-neutralization method

SECONDARY OUTCOMES:
Immunogenicity index-Seroconversion rate of the neutralizing antibody | Day 14 after the full course vaccination
  Neutralizing antibody assay will be performed using the micro-neutralization method. Seroconversion will be defined as a change from seronegative(<1:8) to seropositive(≥1:8), or ≥4 fold increase from baseline
Immunogenicity index-Seropositive rate of the neutralizing antibody | Day 14 after the full course vaccination
  Neutralizing antibody assay will be performed using the micro-neutralization method. Subjects with a antibody titer ≥1:8 will defined as seropositive
Safety index-Incidence of adverse reactions | From the beginning of the vaccination to 28 days after the full course vaccination
  Incidence of adverse reactions from the beginning of the vaccination to 28 days after the full course vaccination
Safety index-Incidence of serious adverse events | From the beginning of the vaccination to 6 months after the full course vaccination
  SAE will be collected throughout the clinical trial

CONTACTS AND LOCATIONS:
Overall Officials: Hongxing Pan, Master, Principal Investigator — Jiangsu Provincial Center for Disease Prevention and Control
Locations (1):
- Dafeng District Center for Disease Prevention and Control, Yancheng, Jiangsu, China